CLINICAL TRIAL: NCT04374643
Title: Descriptive Study of the PSYchological Impact of CONFinement Measures in the General Population : PsyConfPop
Brief Title: Descriptive Study of the PSYchological Impact of CONFinement Measures in the General Population
Acronym: PsyConfPop
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0197
Record Dates: First submitted 2020-04-30; First posted 2020-05-05 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Depression; COVID 19
Keywords: Confinement; Depression; Post traumatic stress; Adults
MeSH Terms: conditions — Depression; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Confined patients: General population
  Interventions: Other: Slef questionnaires fulfilment

INTERVENTIONS:
Other: Slef questionnaires fulfilment — Questionnaires to assess the psychological impact of confinement and its evolution over 6 months

SUMMARY:
Quarantine is an unpleasant experience : separation from loved ones, loss of freedom, uncertainty about infection status, boredom. It may lead to negative mental health consequences and thus the emergence of anxiety and depressive symptoms.

From March 17th, 2020 to May 11th 2002, the French government has implemented national containment measures due to the Covid-19 epidemic.

Although there are data on the psychological impact and experience of quarantine measures in people who have been infected or suspected of being carriers of certain pathogens (e.g. Ebola), there are no data on such impact in the French population and quarantines lasting longer than 21 days. Investigators therefore propose to conduct a human and social sciences study in order to better understand the current situation

DETAILED DESCRIPTION:
The main objective is to describe the psychological state during confinement (and the impact of the confinement) in a sample of the French general population.

Secondary objectives :

* to assess the evolution of psychological health between the period of confinement and post-confinement.
* to identify clinical factors modulating psychological state during confinement

It is expected to highlight :

* a link between the intensity of anxiety symptoms and the number/quality of social contacts
* a reduction of anxiety and depression symptoms in the post-confinement period.
* higher consumption of drugs during the confinement period

Self-questionnaires (Google form format) are sent by mailing lists or social networks to participants in order to complete the assessment of psychological state. A unique identifier is sent in a separate email. These assessments are performed at least once during the confinement period. It is planned to repeat them when the confinement is lifted: 15 days, 3 and 6 months after the lifting of the confinement because of the risk of developing anxiodepressive symptoms, in particular post-traumatic stressors.

ELIGIBILITY:
Inclusion criteria:

- age> 18

Exclusion criteria:

- protective measure (curatorship, guardianship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults who agree to participate by answering the questionnaires
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Depressive Symptomatology | during confinement
  depressive symptomatology with Patient Health Questionnaire : PHQ-9 scale (PHQ 9 higher score, more depressive -> min : 0 max : 27)

SECONDARY OUTCOMES:
Depressive Symptomatology | post-confinement : 15 days, 3 months, 6 months
  depressive symptomatology with Patient Health Questionnaire : PHQ-9 scale (PHQ 9 higher score, more depressive -> min : 0 max : 27)

OTHER OUTCOMES:
Psychological pain | during confinement
  Psychological pain : likert scale (higher score, more psychological pain-> min : 0 max : 10)
sleep | during confinement
  quality of sleep assessed with Insomnia Seveity Index (ISI Insomnia Severity Scale ; higher score, more insomnia -> min : 0 max : 28)
sleep | post-confinement (15 days, 3 months, 6 months)
  quality of sleep assessed with Insomnia Seveity Index (ISI Insomnia Severity Scale ; higher score, more insomnia -> min : 0 max : 28)
anxiety | during confinement
  anxiety intensity assessed by Generalized Anxieety Disorder (GAD 7 Generalized Anxiety Disorder higher score, more anxious -> min : 0 max : 21)
anxiety | post-confinement (15 days, 3 months, 6 months)
  anxiety intensity assessed by Generalized Anxieety Disorder (GAD 7 Generalized Anxiety Disorder higher score, more anxious -> min : 0 max : 21)
psychological pain | post-confinement (15 days, 3 months, 6 months)
  psychological pain : likert scale (higher score, more psychological pain-> min : 0 max : 10)
physical pain | during confinement
  psychological pain : likert scale (higher score, more psychological pain-> min : 0 max : 10)
physical pain | post-confinement (15 days, 3 months, 6 months)
  psychological pain : likert scale higher score, more psychological pain-> min : 0 max : 10)
anger | during confinement
  staxi state scale (STAXI ; State and Trait Anger Expression Inventory : higher score, more anger -> min : 0 max : 50)
anger | post-confinement (15 days, 3 months, 6 months)
  staxi state scale (STAXI ; State and Trait Anger Expression Inventory : higher score, more anger -> min : 0 max : 50)
Stressful Event Impact | during confinement
  Assessed by the Stressful Event Impact Scale - Horowitz (HOROWITZ higher score, more traumatizes -> min : 0 max : 45)
  )
Stressful Event Impact | post-confinement (15 days, 3 months, 6 months)
  Assessed by the Stressful Event Impact Scale - Horowitz (HOROWITZ higher score, more traumatizes -> min : 0 max : 45)
Use of psychotropic drugs | during confinement
  Number of patients declaring an increase of psychotropic drug use
Use of psychotropic drugs | post-confinement (15 days, 3 months, 6 months)
  Number of patients declaring an increase of psychotropic drug use
Tobacco consumption | during confinement
  Number of patients declaring an increase of tobacco consumption
Tobacco consumption | post-confinement (15 days, 3 months, 6 months)
  Number of patients declaring an increase of tobacco consumption
alcohol consumption | post-confinement (15 days, 3 months, 6 months)
  Number of patients declaring an increase of alcohol consumption
alcohol consumption | confinement
  Number of patients declaring an increase of alcohol consumption
Illicit substances consumption | confinement
  Number of patients declaring an increase of illicit substances consumption
Illicit substances consumption | post-confinement (15 days, 3 months, 6 months)
  Number of patients declaring an increase of illicit substances consumption
orientation of life | confinement
  Life Orinetation Test Revised (LOT-R questionnaire): higher score, more optimistic --> min : 0 max : 24
orientation of life | post-confinement (15 days, 3 months, 6 months)
  Life Orinetation Test Revised (LOT-R questionnaire): higher score, more optimistic --> min : 0 max : 24

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Olie, MD PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC